CLINICAL TRIAL: NCT02170766
Title: Bioavailability of BIBR 953 ZW After Single Oral Doses of 12.5, 25, 50 or 100 mg BIBR 1048 MS Film-coated Tablet With and Without Pre-treatment With Pantoprazole to Healthy Subjects. Four Groups, 2-way Crossover, Randomised, Open Trial.
Brief Title: Bioavailability of BIBR 953 ZW in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.15
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Pantoprazole

ARMS (4):
- BIBR 1048 low1 (Experimental): Two treatments of one single dose of BIBR 1048 12.5 mg without or with Pantoprazole
  1. BIBR 1048 12.5 mg without Pantoprazole
  2. BIBR 1048 12.5 mg with 40 mg Pantoprazole (bid)
  Interventions: Drug: BIBR 1048 low1; Drug: Pantoprazole
- BIBR 1048 low2 (Experimental): Two treatments of one single dose of BIBR 1048 25 mg without or with Pantoprazole
  1. BIBR 1048 25 mg without Pantoprazole
  2. BIBR 1048 25 mg with 40 mg Pantoprazole (bid)
  Interventions: Drug: BIBR 1048 low2; Drug: Pantoprazole
- BIBR 1048 medium (Experimental): Two treatments of one single dose of BIBR 1048 50 mg without or with Pantoprazole
  1. BIBR 1048 50 mg without Pantoprazole
  2. BIBR 1048 50 mg with 40 mg Pantoprazole (bid)
  Interventions: Drug: BIBR 1048 medium; Drug: Pantoprazole
- BIBR 1048 high (Experimental): Two treatments of one single dose of BIBR 1048 100 mg without or with Pantoprazole
  1. BIBR 1048 100 mg without Pantoprazole
  2. BIBR 1048 100 mg with 40 mg Pantoprazole (bid)
  Interventions: Drug: BIBR 1048 high; Drug: Pantoprazole

INTERVENTIONS:
Drug: BIBR 1048 low1
  Arms: BIBR 1048 low1
Drug: BIBR 1048 low2
  Arms: BIBR 1048 low2
Drug: BIBR 1048 medium
  Arms: BIBR 1048 medium
Drug: BIBR 1048 high
  Arms: BIBR 1048 high
Drug: Pantoprazole

SUMMARY:
To assess the extend of absorption of 12.5, 25, 50 and 100 mg of BIBR 1048 free base with and without coadministration of 40 mg pantoprazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP and local legislation
* Age ≥ 18 and ≤ 50 years
* Broca ≥ - 20% and ≤ + 20%

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History of current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * Any bleeding disorder including prolonged or habitual bleeding
  * Other hematologic disease
  * Cerebral bleeding (e.g. after a car accident)
  * Commotio cerebri
* Intake of drugs with a long half-life (>24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2000-10; Primary Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
AUC0-inf (Area under the concentration-time curve the time interval from 0 extrapolated to infinity) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
AUC0-tf (Area under the concentration-time curve over the time interval from 0 to the time of the last quantifiable concentration) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug

SECONDARY OUTCOMES:
Cmax (Maximum measured concentration) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
tmax (Time from dosing to the maximum concentration) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
MRTtot (Total mean residence time) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
CLtot/F (Total apparent clearance) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
Vz/F (Apparent volume of distribution) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
λz (terminal elimination rate constant) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
changes in activated partial thromboplastin time (aPTT) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug
changes in international normalized ratio (INR) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 and 48 hours after administration of study drug